CLINICAL TRIAL: NCT03490981
Title: RCT of Brief Cognitive Behavioral Therapy for Chronic Pain
Brief Title: Brief Cognitive Behavioral Therapy for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2741-P; 1I21RX002741-01A1 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: primary care; chronic pain; musculoskeletal pain; cognitive behavioral therapy; integrated primary care
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two arm parallel design: 1) primary care treatment as usual, or 2) primary care treatment as usual and Brief Cognitive Behavioral Therapy for Chronic Pain
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual (TAU) only (Other): Primary care treatment as usual
  Interventions: Other: Treatment as usual (TAU)
- Treatment as usual (TAU) plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) (Experimental): Primary care treatment as usual and Brief CBT-CP
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP)

INTERVENTIONS:
Other: Treatment as usual (TAU) — Participants assigned to TAU will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated.
  Arms: Treatment as usual (TAU) only
Behavioral: Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) — Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6 weeks. Brief CBT-CP session outlines and patient handouts are included in the appendix. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment.
  Arms: Treatment as usual (TAU) plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP)

SUMMARY:
Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) is designed specifically for use in integrated care settings. The first objective of the proposed study is to conduct a pilot randomized controlled trial of Brief CBT-CP compared to primary care treatment as usual to assess feasibility (i.e., recruitment and retention of participants, appropriateness of measures, and assessment of fidelity of service delivery). This trial will also preliminarily assess treatment effectiveness by examining changes in pain-related physical interference, psychological distress, pain intensity, and other related outcomes. Thirty eligible participants will be randomized into either Brief CBT-CP and primary care treatment as usual or primary care treatment as usual only. Eligible Veterans will include those with chronic musculoskeletal pain and pain-related functional impairment identified from primary care. Participants assigned to Brief CBT-CP will receive six sessions of treatment in 30-minute appointments. This intervention will include education and goal setting, activities and pacing, relaxation skills, cognitive coping, and relapse prevention. Assessments will include validated self-report measures that will take place at pre-treatment (baseline), post-treatment, and at 12-week follow-up. The second objective of this study will be to explore patient and provider perceptions of Brief CBT-CP to identify potential modifications that will improve its quality and overall feasibility of delivery in future work. Participants will include up to 12 staff members as well as up to 12 patients who were randomized to Brief CBT-CP. Participants will be interviewed by telephone about key components of the treatment. Participants will comment on protocol and procedures in terms of acceptability (the perception that a treatment is agreeable or that its specific components are satisfactory), appropriateness (the perceived fit or compatibility of the intervention for a given provider or consumer), and feasibility (the extent to which a new treatment can be successfully carried out or is suitable for everyday use). This intervention has clear implications for translation to clinical practice and for improving pain care quality by providing an evidence-based protocol. The potential direct benefit to Veterans includes offering a safe, accessible, non-pharmacological treatment for chronic pain early in the trajectory of care.

DETAILED DESCRIPTION:
We will recruit 30 Veterans from the primary care clinics located at the Buffalo Veterans Affairs medical center in Buffalo, New York. Thirty eligible participants will be randomized in a 1:1 ratio into either (1) Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) plus treatment as usual (TAU) or (2) TAU only. We will engage in recruitment during the second quarter of Year 1 through the end of the first quarter of Year 2. We aim to recruit and enroll 7-8 participants per quarter during that time frame. Post-treatment follow-up will be conducted at eight weeks and at 12 weeks. Two recruitment methods will be used. Veterans with chronic musculoskeletal pain who self-report functional impairment will be referred by their primary care team, in response to a recruitment flyer posted in primary care, or by contacting the principal investigator or study staff directly after hearing of the study by word of mouth or other sources. This approach will be supplemented by a case-finding procedure in which study staff review electronic medical record data to identify potential patients, who will be subsequently contacted by letter and screened by telephone. Following telephone screening, potentially eligible participants will complete a baseline assessment to assess pain and related characteristics as well as remaining exclusion criteria. Those passing baseline measures will be randomized to (1) Brief CBT-CP plus TAU or (2) TAU only. Assignment to Brief CBT-CP will be stratified based on degree of pain interference.

Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6 weeks. Brief CBT-CP session outlines and patient handouts are included in the appendix. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment. Brief CBT-CP will be delivered by a masters-level interventionist either at the medical center or by telephone depending on the preference of the participant.

Participants assigned to TAU only will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated. Participants in TAU only will not receive behavioral intervention from the primary care clinic behavioral health provider.

We will conduct brief interviews with up to 24 purposefully selected participants (i.e., 12 providers and 12 patients). The provider group will include 6 primary care providers and 6 behavioral health providers I providers who staff Veterans Affairs primary care clinics. Interview items are based on implementation constructs relevant for early stage intervention development: acceptability (or agreeableness and satisfaction with treatment components), appropriateness (or perceived fit/compatibility of the intervention), and feasibility (or whether the intervention is suitable for use.) Up to 12 patients who were randomized to Brief CBT-CP will be asked to complete a 30-minute interviews (i.e., telephone or face-to-face, depending on participant preference) following their 12-week assessment (as described in the consent procedures prior to the trial). We will include participants who completed all study procedures but will also attempt to include those who discontinued Brief CBT-CP.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of musculoskeletal pain of three months
* Pain-related functional impairment
* If currently prescribed pain or psychiatric medicine, a stable dose in the last three months (other than over-the-counter medicines)
* Conversant in English
* Established history of Veterans Affairs primary care utilization (i.e., at least one primary care visit in the past year)

Exclusion Criteria:

* Current engagement in psychotherapy or behavioral intervention provided by behavioral medicine services, specialty mental health, or Primary Care Mental Health Integration services for any indication. Note that medication management through these services is not excluded.
* Receiving medical treatments (e.g., surgery, injections) known to impact pain-related outcomes
* Endorsement of imminent suicide risk
* Current substance use problems (i.e., alcohol, opioids, benzodiazepines, or other drugs)
* Unstable psychiatric status (e.g., active psychosis, current mania)
* Diagnosed with major or minor neurocognitive disorder
* Unwilling to have treatment sessions audio recorded

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Beehler, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, New York
Locations (1):
- VA Western New York Healthcare System, Buffalo, New York, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The LDS will contain individual participant data (IPD) that underlie results presented in publications.
Supporting Information: Study Protocol
Time Frame: IPD will be made available for up to three years starting six months after final publication.
Access Criteria: Data will be shared upon completion of a written request and within 90 days of a completed DUA.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual (TAU) Only: Primary care treatment as usual
  TAU: Participants assigned to TAU will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated.
- Treatment as Usual (TAU) Plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP): Primary care treatment as usual and Brief CBT-CP
  Brief CBT-CP: Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6 weeks. Brief CBT-CP session outlines and patient handouts are included in the appendix. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment.
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) Only | Treatment as Usual (TAU) Plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP)
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) Only | Treatment as Usual (TAU) Plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (13.3) | 53.1 (17.3) | 54.1 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
West Haven-Yale Multidimensional Pain Inventory - Interference [Mean (Standard Deviation); unit: units on a scale] — Self-report measure of physical activity interference due to chronic pain. Scores range from 0 to 6, with higher scores indicating higher pain-related interference.
  units on a scale | 3.2 (1.4) | 4.0 (0.8) | 3.6 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: West Haven-Yale Multidimensional Pain Inventory - Interference (WHYMPI-I) to Assess Change at Follow up
Description: The WHYMPI-I is a validated 9-item subscale that evaluates pain-related interference in daily activities and social and occupational functioning. Average scores range from 0 to 6, with higher scores indicating higher pain-related interference.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- TAU Only: Primary care treatment as usual
  TAU: Participants assigned to TAU will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated.
- TAU Plus Brief CBT-CP: Primary care treatment as usual and Brief CBT-CP
  Brief CBT-CP: Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6 weeks. Brief CBT-CP session outlines and patient handouts are included in the appendix. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment.
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
units on a scale | 3.43 (.32) | 3.10 (.33)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .486, ANCOVA; Mean Difference (Final Values) = .33, Standard Error of Mean .47

2. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) to Assess Change at Follow up
Description: This measure is a 9-item measure of depressive symptoms validated for use in primary care. Total scores range from 0 to 27, with higher scores indicating more depression symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 7.35 (.80) | 6.23 (.83)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .342, ANCOVA; Mean Difference (Final Values) = 1.12, Standard Error of Mean 1.16

3. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7) to Assess Change at Follow up
Description: This measure is a 7-item measure of anxiety symptoms validated for use in primary care. Total scores range from 0 to 21, with higher scores indicating more anxiety symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 4.97 (.90) | 5.57 (.94)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .646, ANCOVA; Mean Difference (Final Values) = -.61, Standard Error of Mean 1.31

4. Secondary Outcome: Pain Numeric Rating Scale (NRS) to Assess Change at Follow up
Description: This single-item question asks respondents to rate their average level of pain on an 11-point scale (0-10). Higher scores indicate worse pain.
Time Frame: 12 weeks
Population: N=13 for TAU due to missing NRS data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 13 | 13
score on a scale | 5.37 (.61) | 4.24 (.61)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .205, ANCOVA; Mean Difference (Final Values) = 1.13, Standard Error of Mean .205

5. Secondary Outcome: Pain Self-Efficacy Questionnaire (PSEQ) to Assess Change at Follow up
Description: This validated measure includes 10-items related to pain-related self-efficacy, such as accomplishing goals and becoming more active. Total scores range from 0 to 60, with higher scores indicating greater pain-related self-efficacy.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 37.50 (2.02) | 39.54 (2.10)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .492, ANCOVA; Mean Difference (Final Values) = -2.05, Standard Error of Mean 2.94

6. Secondary Outcome: Pain Catastrophizing Scale (PCS) to Assess Change at Follow up
Description: This validated 13-item measure assesses pain-related cognitions such as pain magnification and perceived helplessness. Total scores range from 0 to 52, with higher scores indicating higher levels of negative pain-related thoughts.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 23.1 (2.6) | 18.8 (2.7)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .272, ANCOVA; Mean Difference (Final Values) = 4.31, Standard Error of Mean 3.84

7. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF) to Assess Change at Follow up
Description: This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains (i.e., physical health, psychological, social relationship, and environment). A total summary score across domains ranges from 24 (minimum) to 120 (maximum), with higher scores indicating greater overall quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 92.1 (3.34) | 92.9 (3.50)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .870, ANCOVA; Mean Difference (Final Values) = -.80, Standard Error of Mean 4.82

8. Secondary Outcome: Ability to Participate in Social Roles and Activities - Short Form (APSRA) to Assess Change at Follow up
Description: This 8-item measure was developed to evaluate one's perceived ability to perform usual social roles and activities. Total scores range from eight to 40, with higher scores indicating better ability to participate in usual activities.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TAU Only | TAU Plus Brief CBT-CP
Number analyzed (Participants) | 14 | 13
score on a scale | 27.76 (1.14) | 26.80 (1.11)
Statistical Analysis 1: Comparison: TAU Only vs TAU Plus Brief CBT-CP; Test type: Superiority; p = .570, ANCOVA; Mean Difference (Final Values) = 0.96, Standard Error of Mean 1.67

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment as Usual (TAU) Only | Treatment as Usual (TAU) Plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (TAU) Only (N=15) | Treatment as Usual (TAU) Plus Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) (N=15)
Stroke symptoms (Vascular disorders) | 1 (1) | 0 (0) — Participant reported to non-VA hospital with possible stroke symptoms. Deemed unrelated to participation in the study.
Back/leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant reported to VA ER with pain in lower back/upper leg. Deemed not related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT03490981/Prot_SAP_000.pdf